CLINICAL TRIAL: NCT06571253
Title: The Comparison of the Efficacy of Online Exercise Prescriptions Delivered Via the Fiziu Digital Physiotherapy Platform and Conventional Paper-Based Exercises in Individuals with Forward Head Posture
Brief Title: Comparison of Online and Paper-Based Exercise Efficacy in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seda GÖZENER CANBÜLBÜL, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: İMU-SEDAGOZENER-003
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This clinical trial employed a randomized controlled design to investigate the effects of a corrective exercise program delivered via the Fiziu Digital Physiotherapy Platform compared to a paper-based exercise program on forward head posture (FHP) in a cohort of adult volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fiziu Digital Physiotherapy Platform Arm (Experimental): Participants in this arm received a 6-week corrective exercise program delivered via the Fiziu Digital Physiotherapy Platform. The program included guided exercise videos, visual and auditory instructions, and automated reminders to ensure adherence. This arm was designed to evaluate the effectiveness of digital exercise delivery in improving forward head posture (FHP).
  Interventions: Behavioral: Digital Exercise Intervention
- Paper-Based Exercise Program Arm (Experimental): Participants in this arm followed a traditional paper-based exercise program for 6 weeks. The program included written instructions and images illustrating the exercises. This arm served as a comparison to evaluate the effectiveness of the traditional exercise delivery method against the digital platform.
  Interventions: Behavioral: Paper-Based Exercise Intervention

INTERVENTIONS:
Behavioral: Digital Exercise Intervention — Participants in this intervention arm used the Fiziu Digital Physiotherapy Platform. This digital platform provided a structured 6-week corrective exercise program through visual and auditory-guided videos. The intervention included interactive features such as reminders and progress tracking to enhance adherence and engagement.
  Arms: Fiziu Digital Physiotherapy Platform Arm
Behavioral: Paper-Based Exercise Intervention — Participants in this intervention arm followed a traditional paper-based exercise program. This included printed exercise instructions and illustrations for a 6-week period. The program was designed to mimic standard physical therapy exercises without digital support.
  Arms: Paper-Based Exercise Program Arm

SUMMARY:
Proper posture is a musculoskeletal balance that minimizes stress on the body and is a key component of orthopedic physical examination. Poor posture, including forward head posture (FHP) and round shoulders, can develop as early as puberty and is exacerbated by prolonged use of smartphones and visual display terminals (VDT), leading to neck and shoulder fatigue and degenerative spine changes. FHP, a common postural issue in the sagittal plane, is associated with thoracic hyperkyphosis and can negatively impact respiratory function by reducing thoracic expansion and lung capacity. FHP also contributes to various musculoskeletal issues, such as temporomandibular disorders, myofascial pain syndrome, and cervicogenic headaches, by increasing biomechanical strain on the posterior neck muscles. Kendall and colleagues describe FHP as a forward positioning of the head, with shortened neck extensors and weakened anterior vertebral neck flexors, leading to muscle fiber damage over time. FHP can be measured using methods like craniovertebral angle (CVA), which is a reliable indicator of FHP severity. Exercise therapy, including strengthening, stretching, and proprioceptive exercises, is recommended to correct FHP and improve postural alignment, potentially enhanced by scapular stabilization exercises. The rise of telehealth presents a promising avenue for treating FHP through accessible and effective telerehabilitation methods. This study aimed to compare the effects of a 6-week home exercise program implemented via the Fiziu digital exercise platform and a traditional paper-based program on FHP and to compare the results between the two groups.

DETAILED DESCRIPTION:
This study aimed to compare the effects of a corrective exercise program delivered via the Fiziu Digital Physiotherapy Platform with those delivered through a paper-based exercise program on volunteers with forward head posture (FHP). The primary objective was to evaluate the impact of these programs on joint range of motion (ROM) and craniocervical angle (CVA) in individuals with FHP and to assess the therapeutic efficacy of a consistent exercise regimen. Additionally, the study sought to determine whether there were differences in outcomes between the digital and paper-based methods, particularly in terms of usability and efficiency.

The study utilized an experimental research design, involving a total of 40 participants, with 20 receiving exercises via the Fiziu platform and 20 following paper-based programs. The intervention lasted six weeks, during which time participants' cervical flexion/extension, lateral flexion (right and left), and rotation (right and left) were measured using a goniometer. The CVA, which represents the angle between the head and the cervical region, was also measured, alongside neck function assessed by the Neck Disability Index (NDI).

Measurements were conducted in a seated position. For cervical flexion and extension, the goniometer's fixed arm was aligned vertically with the floor, with the central point on the C7 vertebra's spinous process. The movable arm was positioned at the external auditory meatus. Participants were instructed to perform maximum flexion and extension movements, and the final angle was recorded. Lateral flexion was measured by placing the goniometer's pivot point on C7, the fixed arm parallel to the floor, and the movable arm aligned with the external occipital protuberance. Participants were asked to bring their ears toward their shoulders, and the final angle was noted. Cervical rotation was measured by placing the goniometer on the vertex of the head, with the fixed arm parallel to the floor and aligned with the nose, and the movable arm following the tip of the nose. Participants rotated their heads to the right and left, and the final angles were recorded.

For CVA measurement, participants maintained a neutral neck position. The goniometer's pivot point was placed on C7, with the fixed arm parallel to the floor and the movable arm aligned with the tragus of the ear. The angle between these two points was recorded.

The NDI was used to measure neck function, which evaluates a person's capacity to perform daily tasks across ten categories: pain intensity, lifting, concentration, reading, headaches, self-care, driving, work, sleep, and recreation. Each category is scored from 0 to 5, with higher scores indicating greater disability.

All measurements were repeated at the end of the study to assess the effectiveness of the interventions.

Inclusion criteria were as follows: participants aged 18-35 years, possessing internet access, and exhibiting a forward head posture (CVA < 50°). Exclusion criteria included: participants under 18 or over 35 years of age, lacking internet access, or having a history of head, neck, or shoulder injuries or surgeries.

The results demonstrated that both the digital and paper-based exercise programs effectively improved joint ROM and CVA in participants with FHP. However, no significant differences were found between the two groups in terms of their impact on CVA. Despite this, the Fiziu Digital Physiotherapy Platform was found to be more user-friendly and efficient compared to the traditional paper-based method, suggesting that digital platforms may offer a practical alternative for delivering therapeutic exercises, especially in telemedicine contexts.

This study fills a gap in the literature by providing insights into the effectiveness of digital exercise platforms for managing FHP, contributing to the broader discussion on the use of new technologies in physical therapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 18-35 years,
* possessing internet access,
* exhibiting a forward head posture (CVA < 50°)

Exclusion Criteria:

* participants under 18 or over 35 years of age,
* lacking internet access,
* having a history of head, neck, and shoulder injuries.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Cervical Joint Range of Motion (ROM) | 6 weeks
  The range of motion of the cervical spine will be measured in flexion, extension, lateral flexion (both right and left), and rotation (both right and left) using a goniometer. These measurements assess improvements in the mobility of the neck, which is directly affected by forward head posture (FHP).
Craniocervical Angle (CVA) | 6 weeks
  The craniocervical angle, defined as the angle between the horizontal line through the external auditory meatus and the line through the 7th cervical vertebra (C7), will be measured using a goniometer. This angle provides an indicator of the severity of FHP.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Gözener Canbülbül, PhD(c), Principal Investigator — İstanbul Medipol Üniversitesi Kavacık Güney Kampüs
Locations (1):
- Istanbul Medipol University, Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaghayegh Fard B, Ahmadi A, Maroufi N, Sarrafzadeh J. Evaluation of forward head posture in sitting and standing positions. Eur Spine J. 2016 Nov;25(11):3577-3582. doi: 10.1007/s00586-015-4254-x. Epub 2015 Oct 17. PMID 26476717
- [Background] Mylonas K, Tsekoura M, Billis E, Aggelopoulos P, Tsepis E, Fousekis K. Reliability and Validity of Non-radiographic Methods of Forward Head Posture Measurement: A Systematic Review. Cureus. 2022 Aug 5;14(8):e27696. doi: 10.7759/cureus.27696. eCollection 2022 Aug. PMID 35935117
- [Background] Jung SI, Lee NK, Kang KW, Kim K, Lee DY. The effect of smartphone usage time on posture and respiratory function. J Phys Ther Sci. 2016 Jan;28(1):186-9. doi: 10.1589/jpts.28.186. Epub 2016 Jan 30. PMID 26957754
- [Background] Szeto GP, Lee R. An ergonomic evaluation comparing desktop, notebook, and subnotebook computers. Arch Phys Med Rehabil. 2002 Apr;83(4):527-32. doi: 10.1053/apmr.2002.30627. PMID 11932856
- [Background] Smithwick W 3rd, Gertner HR Jr, Zuidema GD. Injection of Hypaque (sodium diatrizoate) in the management of abdominal stab wounds. Surg Gynecol Obstet. 1968 Dec;127(6):1215-24. No abstract available. PMID 5727966
- [Background] van der Torn M, Thuma PE, Mabeza GF, Biemba G, Moyo VM, McLaren CE, Brittenham GM, Gordeuk VR. Loading dose of quinine in African children with cerebral malaria. Trans R Soc Trop Med Hyg. 1998 May-Jun;92(3):325-31. doi: 10.1016/s0035-9203(98)91032-x. PMID 9861410
- [Background] Mininni N. [The ethics of appropriateness and the appropriateness of ethics. Comments on a current topic of which we know little and which we discuss even less]. Ital Heart J Suppl. 2000 Apr;1(4):543-6. Italian. PMID 10832142